CLINICAL TRIAL: NCT00525902
Title: An Open-label, Multicenter, Phase II Trial of Adalimumab (Humira) in the Treatment of Refractory Non-infectious Uveitis
Brief Title: Adalimumab (Humira) in the Treatment of Refractory Non-infectious Uveitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Illinois at Chicago (Other); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Eric B. Suhler, Associate Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: e2434
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Results first posted 2012-04-09 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis | interventions — Adalimumab

ARMS (1):
- Adalimumab (Experimental)
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — 40 mg delivered every 2 weeks by subcutaneous injection
  Other Names: Humira

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Adalimumab in uveitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with vision-threatening autoimmune uveitis.
2. Failure to respond to prednisone and at least one other systemic immunosuppressive (such as methotrexate, azathioprine, mycophenolate mofetil, cyclosporine, cyclophosphamide, or chlorambucil), or intolerance to such medications due to side effects.

Exclusion Criteria:

1. Serious concomitant illness that could interfere with the subject's participation in the trial.
2. Previous or current use of cyclophosphamide.
3. Unable or unwilling to undergo multiple injections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric B Suhler, MD, Principal Investigator — Oregon Health and Science University; James T Rosenbaum, MD, Study Director — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adalimumab
Started | 31
10 Weeks | 30
50 Weeks | 12
Completed | 30
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 40.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Endpoint
Description: Improvement in at least one of these criteria without significant worsening in any of them. 1) improvement by 2 or more lines of best-corrected Snellen visual acuity in at least one eye; (2) reduction in dose of systemic corticosteroid or other immunosuppressive therapy by at least 50%; (3) two-step improvement in control of ocular inflammation; and (4) reduction of cystoid macular edema and other inflammatory signs on angiography.
Time Frame: 10 weeks
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 31
participants | 21

2. Primary Outcome: Cumulative Endpoint
Description: as for outcome 1
Time Frame: 50 Weeks
Population: Participants characterized as clinical responders at 10 weeks were allowed to continue in the study.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 21
participants | 12

ADVERSE EVENTS:
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 6/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=31)
Hypoglycemic Coma (Blood and lymphatic system disorders) | 1 (1)
Stroke (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=31)
Headache (General disorders) | 3 (3)
Joint pain (General disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
2 had to discontinue for methodologic reasons (pregnancy, loss to follow up wk 42), leading to their classification as failures. As a three-center study, differences between the study population are possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes